CLINICAL TRIAL: NCT05947682
Title: Manufacturing of Allogeneic Adipose Tissue-derived Mesenchymal Stromal Cells for Treatment of Severe Systemic Sclerosis
Acronym: Pre_MSC-AT-SSc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230376
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Mesenchymal Stromal Cell; Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults who are planned to undergo plastic surgery (Other): Adults who are planned to undergo plastic surgery for abdominal liposuction or lipoaspiration under general anaesthetic for their own care and who are voluntary for fat donation to contribute to the study
  Interventions: Other: Adipose tissue harvesting

INTERVENTIONS:
Other: Adipose tissue harvesting — Adipose tissue harvesting (40-60g) during the abdominal liposuction or lipoaspiration under general anaesthesia which is performed according to usual care

SUMMARY:
Mesenchymal stromal cells (MSC) are multipotent cells which carry immunomodulatory, pro-angiogenic and anti-fibrotic properties, that can target Systemic Sclerosis (SSc) pathogenesis and its clinical manifestations. The increasing use of MSC, harvested from bone marrow (MSC(M)), adipose tissue (MSC(AT)), or umbilical cord (MSC(UC)) in a variety of indications, provides consistent evidence supporting their safety in humans. The efficacy of MSC(M) intravenous (IV) injection for treating acute graft versus host disease led to their marketing approval in 2012 and MSC(AT) (Alofisel) were approved for severe Crohn's fistula in 2018.

MSC represent a promising therapeutic approach for SSc. We previously a) showed disease-specific abnormalities in MSC(M) from SSc patients, providing strong rationale to use allogeneic MSC to treat SSc patients, b) completed the first phase I/II dose escalation trial using allogenic MSC(M) infusion in 20 severe SSc patients (ClinicalTrials.gov: NCT02213705, PHRC AOM 11-250) with no safety issues, significant improvement in skin fibrosis at 3 to 6 months after infusion which appeared lower thereafter, thereby supporting the need for repeated infusions.

In vitro, experimental and clinical studies suggest that MSC properties vary according to their tissue of origin/source. We demonstrated that compared to MSC(M), MSC(AT) are easier to harvest and display higher proliferative capability before entering senescence, higher genetic stability, and superior immunosuppressive properties.

The objective of the present research is the successful production of allogeneic MSC(AT) derived from selected healthy donors, with adequate phenotypic criteria according to the International Society for Cell & Gene Therapy.

Considering the above rationale, these MSC(AT) will subsequently be used in a Phase I/II randomized clinical trial testing allogeneic MSC(AT) systemic infusion for treatment of severe systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 55 years
* BMI <30
* Non-smoker
* Admission for a pre-scheduled plastic surgery intervention liposuction or lipo-aspiration in the abdominal wall under general anesthesia
* Written consent
* Affiliated to a social security

Exclusion Criteria:

* Weight < 50 kg
* Positive viral serology : Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV), Hepatitis E Virus (HEV), syphilis, Human T Lymphotropic virus (HTLV), active infection with IgM+ for toxoplasmosis, Epsiten Barr Virus (EBV), Cytomegalovirus (CMV)
* Active generalized infection (viral, parasitic, tuberculosis, leprosy...)
* Significant comorbidities according to donor health history or existing risk factors for viral infections within the past 12 months:

  * Multiple sexual partners between the donor or his or her usual partner
  * Intravenous addiction to the donor or regular partner
  * Accident of exposure to blood or derivatives suspected of being contaminated
* Uncontrolled hypertension
* Human dura mater transplant
* Surgical history of the central nervous system
* Dementia or neurological disease that may evoke subacute spongiform encephalopathy
* Family history as part of subacute spongiform encephalopathy
* Hematological malignancies
* Active or any past history of cancer
* History of chemotherapy or irradiation
* Systemic or autoimmune disease
* Multiple adenopathy, splenomegaly, hepatomegaly
* Icterus
* Haemophilia
* Known insulin-dependent diabetes
* Treatment with extractive pituitary hormones (including growth hormones)
* Steroids therapy (for more than 5 days) in the past 3 months
* Lithium treatment
* Pregnancy
* Deprived of freedom

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Production of at least 3 batches of MSC(AT) derived from donors adipose tissue | Up to 2 months

SECONDARY OUTCOMES:
Percentage of viability | Up to 2 months
Percentage of CD73+ cells | Up to 2 months
Percentage of CD90+ cells | Up to 2 months
Percentage of CD105+ cells | Up to 2 months
Percentage of expression of HLA-DR | Up to 2 months